CLINICAL TRIAL: NCT03174080
Title: PET MRI for Evaluation of Knee Osteoarthritis in Patients With Bilateral Knee OA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, david groshar, Pro. David Groshar, Assuta Medical Center
Other Study IDs: Assuta MC
Record Dates: First submitted 2016-12-28; First posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Knee Osteoarthritis
Keywords: Positron-Emission; PET Scan Tomography
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — without biospecimen
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: FDG (glucose labeled isotope of fluorine) — Patients will receive an intravenous injection of 2-5mCi of 18F-FDG prior to PET MRI

SUMMARY:
Osteoarthritis (Osteoarthritis) of the knee is a high prevalence in the population of people aged 60 years and over, when in some cases does not cause any discomfort or pain, and therefore not diagnosed. In addition, Radio graphic findings of the knee not fully compatible with the patient's symptoms, which resulted in errors in the interpretation and diagnosis.

In this study, patients who suffer from two knees or unilateral pain, will take part. Participants will undergo a clinical examination, including evaluation of symptoms by an orthopedist and an X-ray imaging, which are part of the currently accepted medical diagnosis.

Patients will perform PET-MRI test in order to assess whether PET MRI is a more efficient tool for active knee osteoarthritis diagnosis.

DETAILED DESCRIPTION:
Knee Osteoarthritis has high incidence in the population over 60 years reaching a rate of 10% in several studies. However, not all arthritic knee joints are actively causing patient discomfort or pain. There is only a limited correlation between patient radio graphs and symptoms leading to high rates of false positive and false negative of knee OA. Consequently, patients may have bilateral knee arthritis when the more arthritic knee per x-ray is less symptomatic. On the other hand knee MRI and bone scan maybe oversensitive for diagnosis knee arthritis with a high rate of false positive.

The purpose of this study is to examine the value of PET MRI as a tool for accurate diagnosis of active knee osteoarthritis.

The hypothesis is that using PET MRI of both knees may correlate better than radio graphs or MRI by themselves to patient symptoms .

The study will consist of 150 patients with bilateral or unilateral knee pain with one of the knees having more symptoms than the other. The study physicians who perform the PET MRI will be blinded to the patient symptoms and will record their findings and which knee is more symptomatic and along which pattern

Enrollment:

* All patients that are sent for knee MRI
* Patients over the age of 50 years old
* All patients will sign an informed consent for the study prior to the PET MRI
* Unilateral or Bilateral knee pain
* All patients were ambulatory preoperative, using no more then a single cane
* All patients had prior Weight Bearing AP x-rays and Lateral radiography The patients will be fill in SF-36 and WOMAC and VAS scores along prior to their examination.

All patients will have an orthopedic assessment of their symptoms prior to their PET MRI.

Participants will carry out a PET-MR imaging. PET involves injecting FDG (glucose labeled isotope of fluorine) intravenously at a dose of 2.5 mci . After a wait of about 40 minutes will be performed PET MR lasting up to 40 minutes.

All findings will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* All patients that are sent for knee MRI
* Patients over the age of 50 years old
* All patients will sign an informed consent for the study prior to the PET MRI
* Unilateral or Bilateral knee pain
* All patients were ambulatory pre-operatively, using no more then a single cane
* All patients had prior Weight Bearing AP x-rays and Lateral Radiogrphs

Exclusion Criteria:

1. Non ambulatory patients
2. History of knee arthroscopy or other surgery 1 year before the MRI
3. Bone scan performed in the past 3 months prior to the PET MRI
4. Clastrophobia

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will consist of 150 patients with bilateral or uniltarel knee pain with one of the knees having more symptoms than the other.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-07-16 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
correlation between SUV to clinical evaluation | 3 months - 1 year
  correlation between SUV PET vs. WOMAC and VAS pain scores.

IPD SHARING:
Plan to Share IPD: No
IPD